CLINICAL TRIAL: NCT06799871
Title: Retrospective Single Cohort Mono-center Study on Trends in Implant Stability Measured by RFA
Brief Title: RFA R-Evolution: a New Protocol to Avoid Implant Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Daniele Moretto (Other)
Responsible Party: Sponsor-Investigator, Daniele Moretto, Dr, Odontoiatri Associati, Bologna
Organization: Odontoiatri Associati, Bologna (Other)
Other Study IDs: 2024-1806
Record Dates: First submitted 2024-12-12; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-12

CONDITIONS: Dental Implants
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Dental implant — There is no intervention in the study. The participants have already received dental implant treatment and data will be collected retrospectively regarding the procedure

SUMMARY:
The main objective of this study is to assess the impact of confounding factors such as jaw, implant position, indication, smoking status, implant dimension, and medical history on RFA trends. In addition, this study aims to explore correlations of RFA trend, with the goal of using ISQ trends as an indicator for treatment protocol decisions (e.g. time of loading). Participants have already received dental implant as per clinic's standard protocol. Information regarding Implant Stability Quotient (ISQ) measurements performed at any time point until 1-year follow-up will be collected. The principal investigator protocol regarding the use of ISQ measure to define time of implant loading will also be assessed. Only participants followed up at least until one year after implant placement will be included in the data collection.

DETAILED DESCRIPTION:
This single-center retrospective study includes all consecutive participants treated since October 2021 for single or multiple edentulous sites (either healed or extracted). Only participants with a 1-year follow-up visit and RFA measurements at three or more time-points are included.

Participants will be consecutively included provided they meet all of the inclusion criteria and none of the exclusion criteria. As the data is anonymized, participants will not be contacted for consent.

Any additional post-hoc exclusion of participants will be thoroughly documented.

The primary endpoint of the study is:

-Occurrence of RFA trends (3 consecutive increasing or stable RFA values vs 3 consecutive decreasing RFA values)

Secondary endpoints:

* Implant treatment success (implant loaded functionally) after 1 year of implant placement
* Change in prosthetic protocol (3 months to definitive prosthesis placement in maxilla, 2 months in mandible) due to ISQ trend

Participants have already received dental implant(s) at surgery visit. Implant Stability Quotient (ISQ) was assessed after implant placement. Depending on the trends in ISQ, implants were loaded with provisional and the final prosthesis and followed up at least until 1 year after surgery.

Data collection methods Data will be collected by automatic extraction from the clinic's patient management system and will for statistical analysis.

Implant is considered survived if it is in-situ. Implant treatment success is defined as implant loaded functionally.

Demographic data will be collected in the automatic extraction of the data and used to access participant's eligibility to partake in the study.

Any relevant medical history of participants will be collected in the automatic extraction as well. Demographic and medical history data will also be part of the data analysis.

At interim and 1-year follow-up visits, prosthetic parameters will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Participant received implant treatment NobelReplace, NobelActive or NobelParallel implants on or after October 2021 (with TiUnite or TiUltra surfaces)
* Participant was at least 18 years old at the time of surgery
* Participant attended a follow-up visit at least 1-year after surgery
* Implant stability was assessed by means of RFA at a minimum of three time-points

Exclusion Criteria:

* 1-year follow-up data not available
* Subject received major guided bone regeneration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 100 consecutive subjects treated with the RFA-trend protocol since October 2021 are included. To ensure sufficient sampling of underrepresented indications and due to the novelty of this decision-making protocol, adaptive sample size determination will be used.
  Participant received implant treatment NobelReplace, NobelActive or NobelParallel implants on or after October 2021 (with TiUnite or TiUltra surfaces)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Resonance frequency analysis (RFA) trends | From implant insertion until definitive prosthesis delivery (3 months after implant insertion). Time duration 3 months
  Occurrence of Resonance frequency analysis trends (3 consecutive increasing or stable implant stability quotient (ISQ) values vs 3 consecutive decreasing ISQ values)

SECONDARY OUTCOMES:
Implant treatment success | Until 1 year after implant insertion
  Implant loaded functionally after 1 year of implant placement
Change in prosthetic protocol | Until 1 year after implant insertion
  3 months to definitive prosthesis placement in maxilla, 2 months in mandible due to ISQ trend

IPD SHARING:
Plan to Share IPD: No